CLINICAL TRIAL: NCT02712034
Title: Impact on Opioid Use of Bundling Medication-assisted Treatment With mHealth
Acronym: Bundling
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Stanley Street Treatment and Resources (SSTAR) (Unknown); Gosnold on Cape Cod (Unknown); ARC Community Services, Inc. (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2015-1418; 1R01DA040449-01 (NIH); A195010 (Other: UW Madison); INDUSTRIAL ENGR\CHESS PROG (Other: UW Madison)
Record Dates: First submitted 2016-03-14; First posted 2016-03-17 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Opioid Use Disorder
Keywords: Medication-assisted treatment (MAT); Buprenorphine; Methadone; Naltrexone
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Medication-assisted treatment (MAT) (Placebo Comparator): Patients will receive standard medication-assisted treatment (MAT) as prescribed by their health care provider.
  Interventions: Other: MAT
- MAT + A-CHESS (Experimental): Patients in the MAT + A-CHESS arm will receive MAT as described plus the A-CHESS recovery support system via a smartphone.
  Interventions: Behavioral: MAT + A-CHESS

INTERVENTIONS:
Behavioral: MAT + A-CHESS — Subjects randomized to MAT + A-CHESS will receive MAT plus the A-CHESS recovery support system which provides:
  1. Self-directed, interactive modules that teach basic recovery support, harm-reduction, and psychosocial functioning skills.
  2. The latest information about addiction and recovery support, monitoring prompts, and peer and family support.
  3. Advice on where to go for help and on how to make the best use of health and human services; and
  4. A way to talk with experts in the area of addiction and other study participants by sending anonymous messages in the A-CHESS discussion groups.
  5. A way to keep your health care team up to date through reports based on information entered into A-CHESS (i.e. alcohol and drug use, depression, MAT side effects).
  Arms: MAT + A-CHESS
Other: MAT — Patients will receive treatment consisting of a recovery plan, appropriate pharmacology, routine urine screens, and regularly scheduled behavioral interventions, such as monthly group counseling sessions or sessions with a recovery coach. "Appropriate pharmacology" may include methadone; naltrexone; buprenorphine; and in the case of overdose, naloxone; and other medications and combinations of medications as part of the patient's standard clinical care.
  Arms: Medication-assisted treatment (MAT)

SUMMARY:
The primary aim of this study is to measure and explain the impact on long-term opioid use when medication-assisted treatment (MAT) is bundled with an evidence-based mobile-health system (A-CHESS).

ELIGIBILITY:
Inclusion Criteria:

1. are 18+ years old;
2. meet criteria for opioid use disorders of at least moderate severity (4 or 5 DSM-V criteria);
3. Are currently taking medication-assisted treatment (MAT) as part of their standard clinical care;
4. have no acute medical problem requiring immediate inpatient treatment;
5. have no history of psychotic disorders, though those with other co-morbid psychopathology (mood disorders, anxiety, other substance use disorders) will be eligible;
6. are willing to participate in a randomized clinical trial;
7. provide the name, verified telephone number, and address of at least 2 contacts willing to help locate the patient, if necessary, during follow-up;
8. are able to read and write in English;
9. are not pregnant;
10. are willing to share health-related data with primary care clinicians; and
11. are, at study intake, abstinent from opioids for at least 1 week and no longer than 2 months, except for medications used to treat the disorder (e.g., methadone).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 417 (Actual)
Dates: Start 2016-04-21 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Opioid use | 24 months
  Detect the difference in illicit opioid use between patients who have MAT + A-CHESS vs. MAT alone.

CONTACTS AND LOCATIONS:
Overall Officials: David H Gustafson, PhD, Principal Investigator — UW Madison
Locations (1):
- Access Community Health Centers, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hochstatter KR, Gustafson DH Sr, Landucci G, Pe-Romashko K, Cody O, Maus A, Shah DV, Westergaard RP. Effect of an mHealth Intervention on Hepatitis C Testing Uptake Among People With Opioid Use Disorder: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2021 Feb 22;9(2):e23080. doi: 10.2196/23080. PMID 33616545
- [Derived] Hochstatter KR, Gustafson DH Sr, Landucci G, Pe-Romashko K, Maus A, Shah DV, Taylor QA, Gill EK, Miller R, Krechel S, Westergaard RP. A Mobile Health Intervention to Improve Hepatitis C Outcomes Among People With Opioid Use Disorder: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Aug 1;8(8):e12620. doi: 10.2196/12620. PMID 31373273
- [Derived] Gustafson DH Sr, Landucci G, McTavish F, Kornfield R, Johnson RA, Mares ML, Westergaard RP, Quanbeck A, Alagoz E, Pe-Romashko K, Thomas C, Shah D. The effect of bundling medication-assisted treatment for opioid addiction with mHealth: study protocol for a randomized clinical trial. Trials. 2016 Dec 12;17(1):592. doi: 10.1186/s13063-016-1726-1. PMID 27955689